CLINICAL TRIAL: NCT03583944
Title: Post Marketing Trial (Phase IV) on the Safety, Tolerability And Efficacy of Eribulin Mesylate in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study to Evaluate Safety, Tolerability and Efficacy of Eribulin Mesylate in Treating Adult Females With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-M065-401
Record Dates: First submitted 2018-06-20; First posted 2018-07-12 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2018-07

CONDITIONS: Breast Neoplasms
Keywords: E7389; Tumors, Breast; Breast Cancer; Breast Carcinoma; Neoplasms, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eribulin Mesylate 1.23 mg (Experimental): Participants will receive eribulin mesylate 1.23 mg intravenous (IV) infusion, given over 2 - 5 minutes on Days 1 and 8 of 21 days cycle for a total of 6 cycles.
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate IV infusion.
  Other Names: Halaven

SUMMARY:
The purpose of this study is to evaluate clinical and laboratory safety of eribulin mesylate in treating participants with locally advanced or metastatic breast cancer, who have progressed after at least one regimen of chemotherapy which has included anthracycline and taxane therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with locally advanced or metastatic breast cancer.
2. Participants must have progressed after at least after at least one chemotherapeutic regimen for advanced disease. Prior therapy should have included an Anthracycline and a Taxane unless participants who are not suitable for these treatments.
3. Participants must have documented disease progression within or on 6 months from their last anti-cancer therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 2.
5. Participants must have normal organ and marrow function as defined below:

   * Absolute neutrophil count greater than (>) 1,500 per microliter (/mcL)
   * Hemoglobin >10.0 gram per deciliter (g/dL)
   * Platelets >100,000/mcl
   * Serum total bilirubin less than (<) 1.5*upper limit of normal (ULN)
   * Serum aspartate aminotransferase (AST) (Serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (Serum glutamic pyruvic transaminase [SGPT]) <3*ULN or <5*ULN in the presence of liver metastases
   * Serum creatinine <1.5 mg/dL.
6. Females in reproductive age willing to follow adequate barrier contraceptive measures during the conduct of study.

Exclusion Criteria:

1. Hypersensitivity to the active substance or any of the excipients.
2. Participants who have received chemotherapy, radiation, or biological therapy within two weeks, or hormonal therapy within one week before study treatment start, or any investigational drug within four weeks before study treatment start.
3. Participants receiving any other investigational agents.
4. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, recent myocardial infarction, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, or other comorbid condition that investigator believes may compromise participant's condition.
5. Participants requiring concurrent anti-cancer therapy during the study period.
6. Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline up to 30 days after last dose of study drug or at discontinuation (approximately up to 17 months)
  Clinical Safety will be assessed by recording the adverse events (AEs) and serious AEs (SAEs) observed during the study period and its relation to the study medication. AE is defined as any untoward medical occurrence in a participant administered a treatment of medicinal product. An SAE is any untoward medical occurrence that at any dose results in death, results in life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity or results in a congenital anomaly/birth defect.
Number of Participants with TEAEs Related to Laboratory Parameters | Baseline up to 30 days after last dose of study drug or at discontinuation (approximately up to 17 months)
  AE is defined as any untoward medical occurrence in a participant administered a treatment of medicinal product. An SAE is any untoward medical occurrence that at any dose results in death, results in life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity or results in a congenital anomaly/birth defect. TEAEs are defined as those events that started on or after the date and time of administration of the first dose of study drug and those events that were present prior to the administration of the first dose of study drug and increased in severity during the study.

SECONDARY OUTCOMES:
Objective Tumor Response | Baseline to first date of documented CR, PR, SD, or PD, up to end of study treatment (approximately up to 17 months)
  Radiological confirmation of objective response rate (ORR) will be assessed by the Response Evaluation Criteria in Solid Tumors(RECIST)criteria version 1.1. The response would be assessed based on the four response parameters -complete response(CR), partial response(PR), stable disease(SD), progressive disease(PD).CR is defined as disappearance of all target lesions. PR is seen when there is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameters. When there is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of longest diameters since the treatment started then, the response is evaluated as SD.PD is seen when there is at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions.
Objective Response Rate (ORR) | Baseline to first date of documented CR, PR, SD, or PD, up to end of study treatment (approximately up to 17 months)
  ORR measures the response rate using the formula - CR+PR/ (number of eligible participants)*100. CR is defined as disappearance of all target lesions. PR is seen when there is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Eisai Inc.
Locations (18):
- India (18):
  - HEMATO-ONCOLOGY CLINIC Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - HealthCare Global Enterprises Ltd, Bangalore, Karnataka
  - Srinivasam Cancer Care Multispecialty Hospitals India Pvt Ltd, Bangalore, Karnataka
  - KR Hospital Mysore Medical College, Mysore, Karnataka
  - Tata Memorial Hospital Department of Oncology, Mumbai, Maharashtra
  - HCG NCHRI Cancer Centre, Nagpur, Maharashtra
  - Lokmanya Hospital, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Deep Hospital, Ludhiana, Punjab
  - Sawai Man Singh Hospital, Jaipur, Rajasthan
  - MNJ Institute of Oncology and Regional Cancer Centre, Hyderabad, Telangana
  - J.K.Cancer Institute, Kanpur, Uttar Pradesh
  - King George's Medical University,(Erstwhile Chhatrapati Shahuji Maharaj Medical University), Lucknow, Uttar Pradesh
  - Ajanta Research Centre, Ajanta Hospital & IVF Centre, Lucknow, Uttar Pradesh
  - Nilratan Sircar Medical College and Hospital, Kolkata, West Bengal
  - Netaji Subhash Chandra Bose Cancer Institute, Kolkata, West Bengal
  - IPGME&R S.S.K.M Hospital, Kolkata, West Bengal